CLINICAL TRIAL: NCT01972620
Title: Prospective Randomized Controlled Trial (PRCT) Comparing Standard Analgesia With Multi-modal Targeted Operative and Port-Site Local Anesthesia for Post-Operative Pain Management in Elective Laparoscopic Cholecystectomy (LapChole)
Brief Title: RCT: Multi-modal Analgesia for Laparoscopic Cholecystectomy
Acronym: LapChole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinicki Centar Vojvodine (Other)
Responsible Party: Principal Investigator, Radovan Veljkovic, M.D., Ph.D., MD, PhD, ass. prof, Klinicki Centar Vojvodine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00-01/515
Record Dates: First submitted 2013-10-16; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Gallstones; Cholelithiasis; Pain
Keywords: gallstones; cholelithiasis; cholecystectomy, laparoscopic; pain
MeSH Terms: conditions — Gallstones; Cholelithiasis; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-modal analgesia (Active Comparator): Thirty-one patients were enrolled in this arm. Standard analgesia according to institutional standard and 50:50 mixture of normal saline (8 ml) and 0.5% Bupivacaine was prepared within a 20 ml syringe (Total volume = 16 ml; Final concentration = 0.25%). Following delivery of the gallbladder specimen 8 ml of 0.25% bupivacaine solution was sprayed onto the cystic plate (gallbladder fossa) with a spinal needle advanced under direct laparoscopic vision via a 5mm right subcostal laparoscopic port. The anesthetic solution was sprayed at an operating distance from the cystic plate of ~ 2 cm. Following evacuation of the pneumoperitoneum, the remaining 8 ml of 0.25% Bupivacaine was infiltrated subcutaneously at each of the 4 laparoscopic port sites (2 ml per port site) prior sutured closure.
  Interventions: Drug: Bupivacaine
- Control (No Intervention): Thirty-two patients were enrolled in this arm. They received standard analgesia according to institutional standard of practice consisted of non-narcotic analgesia with narcotic analgesic rescue after laparoscopic cholecystectomy.

INTERVENTIONS:
Drug: Bupivacaine — A 50:50 mixture of normal saline (8 ml) and 0.5% Bupivacaine was prepared within a 20 ml syringe (Total volume 16 ml; Final concentration = 0.25%). Following delivery of the gallbladder specimen in the Multi-modal analgesia group, 8 ml of 0.25% bupivacaine solution was sprayed onto the cystic plate (gallbladder fossa) with a spinal needle advanced under direct laparoscopic vision via a 5mm right subcostal laparoscopic port. The anesthetic solution was sprayed at an operating distance from the cystic plate of ~ 2 cm. Following evacuation of the pneumoperitoneum, again within the Multi-modal analgesia group, the remaining 8 ml of 0.25% Bupivacaine was infiltrated subcutaneously at each of the four laparoscopic port sites (2 ml per port site) prior to standard sutured closure of each incision
  Other Names: Marcaine; Bupivacaine HCL
  Arms: Multi-modal analgesia

SUMMARY:
Analgesic efficacy of multi-modal analgesia is superior to standard analgesia for patients undergoing elective laparoscopic cholecystectomy for symptomatic cholelithiasis. Topical cystic plate and port-site incision 0.25% bupivacaine significantly reduces pain after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Background: Peri-portal nerve stimulation has recently been suggested as a mechanism for pain after laparoscopic cholecystectomy (LapChole). We therefore conducted a PRCT to evaluate whether somatovisceral pain blockade reduces pain after LapChole.

Hypothesis:Analgesic efficacy of multi-modal analgesia is superior to standard analgesia for patients undergoing elective LapChole for symptomatic cholelithiasis. Specifically, topical cystic plate and port-site infiltrationwith0.25% bupivacaine significantly reduces pain after LapChole.

Design: Single-blinded PRCT Setting: Academic medical centers Patients and Methods: Between February and May 2010 we randomly assigned 63 patients with symptomatic cholelithiasis in a 1:1 ratio to institutional standard non-opioid/opioid analgesic combinations (n=32), and institutional standard analgesia plus topical 0.25%bupivacaine spray onto the cystic plate and local 0.25% bupivacaine port-site injection,post-LapChole (n=31). Primary endpoint was patient-reported pain 1, 4, 6, 12, and 24 hours, and 1 week post-LapCholeusing the Visual Acuity Score (VAS, 0-10).

Results: Study groups were comparable clinicopathologically. There were no study-procedure-associated adverse events. A statistically significant reduction in mean pain score was apparent in patients receiving multi-modal analgesia at all early (1-6 hours) post-operative time points and at one week following LapChole(p<0.05).

Conclusion: This PRCT shows significantly improved pain reduction with somatovisceral pain blockade than institutional standard analgesic combinations following LapChole for symptomatic cholelithiasis. For centers not utilizing adjunctive local anesthetic for this operation, this multi-modal analgesic approach can improve patient comfort during recovery.This approach serves as the basis for a planned 4-arm PRCT designed to provide further insights into the role of local anesthetics in multi-modal operative site analgesia.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic cholelithiasis undergo elective laparoscopic cholecystectomy
* non - pregnant women
* 18 years or older

Exclusion Criteria:

* undergoing urgent cholecystectomy
* patients operated on for indications other than symptomatic cholelithiasisT
* those having conversion from laparoscopic to open cholecystectomy
* those that withdrew from the study for any reason before the end of the required 7-day follow up (including those that died during that period)
* those with incomplete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Visual Scale Pain VAS | from 0 to 7 postoperative days
  The primary endpoint was patient-reported pain 1, 4, 6, 12, and 24 hours, and 7 days following laparoscopic cholecystectomy using the Visual Acuity Score (VAS, 0-10).

SECONDARY OUTCOMES:
nausea | from 0 to 6 hours post-operatively
  Surgical outcome data recorded prospectively also included severity of post-operative nausea (measured VAS, 0 none and 10 worst state) on one and six hours post-operatively.

OTHER OUTCOMES:
mobility | from 0 to 7 postoperative days
  Surgical outcome data recorded prospectively also included hospital stay (days), impairment of mobility [measured with VAS, 0 is worst and 10 optimal mobility (pre-operative baseline)] one and seven days post-operatively,

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Veljkovic, MD, PhD, Principal Investigator — Clinical Centre of Vojvodina
Locations (1):
- Klinicki Centar Vojvodine, Novi Sad, Vojvodina, Serbia

REFERENCES:
- [Result] Verma GR, Lyngdoh TS, Kaman L, Bala I. Placement of 0.5% bupivacaine-soaked Surgicel in the gallbladder bed is effective for pain after laparoscopic cholecystectomy. Surg Endosc. 2006 Oct;20(10):1560-4. doi: 10.1007/s00464-005-0284-5. Epub 2006 Aug 1. PMID 16897291
- [Result] Boddy AP, Mehta S, Rhodes M. The effect of intraperitoneal local anesthesia in laparoscopic cholecystectomy: a systematic review and meta-analysis. Anesth Analg. 2006 Sep;103(3):682-8. doi: 10.1213/01.ane.0000226268.06279.5a. PMID 16931681
- [Result] Mitra S, Khandelwal P, Roberts K, Kumar S, Vadivelu N. Pain relief in laparoscopic cholecystectomy--a review of the current options. Pain Pract. 2012 Jul;12(6):485-96. doi: 10.1111/j.1533-2500.2011.00513.x. Epub 2011 Oct 19. PMID 22008277
- [Result] Gupta A. Local anaesthesia for pain relief after laparoscopic cholecystectomy--a systematic review. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):275-92. doi: 10.1016/j.bpa.2004.12.007. PMID 15966498